CLINICAL TRIAL: NCT06025305
Title: Development and Validation of Multi-scale Deep Neural Network-Based CT Intelligent Diagnosis System for Coronary Vulnerable Plaques: A Chinese Multicenter Study
Brief Title: Identifying Vulnerable CoronAry PLaqUes With Artificial IntElligence-assisted CT Angiography
Acronym: VALUE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang longjiang,MD, Director, Head of Radiology, Principal Investigator, Jinling Hospital, China
Other Study IDs: 2023DZKY-058-01
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Plaque, Atherosclerotic
Keywords: artificial intelligence; coronary CT angiography; vulnerable plaque
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent coronary CT angiography and intravascular ultrasound within 3 months
  Interventions: Diagnostic Test: Intravascular imaging test
- Patients who underwent coronary CT angiography and optical coherence tomography within 3 months
  Interventions: Diagnostic Test: Intravascular imaging test

INTERVENTIONS:
Diagnostic Test: Intravascular imaging test — Coronary artery disease patients first underwent CCTA and then intravascular imaging test within 3 months

SUMMARY:
The goal of this observational study is to develop an automatic whole-process AI model to detect, quantify, and characterize plaques using coronary CT angiography in coronary artery disease patients. The main questions it aims to answer are:

1. Whether the AI model enables to detect and quantify coronary plaques compared with intravascular ultrasound or expert readers;
2. Whether the AI model enables to identify vulnerable plaques using intravascular ultrasound or optical coherence tomography as the reference standard.
3. Whether the AI model enables to predict future adverse cardiac events in a large cohort of 10,000 patients with non-obstructive CAD.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains the leading cause of death worldwide. Atherosclerotic plaques play a pivotal role in CAD-related patient mortality. Thus, the detection, quantification, and characterization of coronary plaques are clinically significant for early prevention and interventions for CAD.

Coronary CT angiography (CCTA) has emerged as a robust noninvasive tool for the evaluation of CAD. In clinical practice, the coronary plaque assessment is performed by a time-consuming manual process dependent on the clinician's experience and subjective visual interpretation. With the development of artificial intelligence, many automatic computer-aided methods have been proposed to post-process the CCTA images. However, previously proposed algorithms of plaque evaluation were not developed based on intravascular ultrasound (IVUS) or optical coherence tomography (OCT), which were regarded as the gold reference for plaque evaluation. Thus, we aimed to develop a deep learning model in a whole-process automatic and intelligent system on CCTA to detect, quantify, and characterize plaques using IVUS or OCT as reference standard. Then we will work on the validation in different clinical scenarios: (1) Validation of the accuracy of the new deep learning model; (2) Prognosis of the model in different populations with CAD.

The main questions it aims to answer are:

1. Whether the AI model enables to detect and quantify coronary plaques compared with intravascular ultrasound or expert readers;
2. Whether the AI model enables to identify vulnerable plaques using IVUS or OCT as the reference standard.
3. Whether the AI model enables to predict future adverse cardiac events in a large cohort of 10,000 patients with non-obstructive coronary artery disease (China CT-FFR study 2).

ELIGIBILITY:
Inclusion Criteria:

* Intravascular imaging (including intravascular ultrasound or optical coherence tomography) was performed within 3 months after CCTA;
* No change in medications or clinical symptoms during CCTA and intravascular imaging examinations;
* Coronary artery diameter stenosis of 30% to 90% on invasive coronary imaging.

Exclusion Criteria:

* Image quality of CCTA or intravascular US was inadequate to analyze;
* Intravascular imaging was performed after percutaneous coronary intervention (PCI) or pre-dilation of the target lesions;
* Lesions could not be co-registered between CCTA and intravascular US;
* Missing CCTA or intravascular US data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients who first underwent CCTA and then Intravascular imaging in China
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of AI-assisted coronary CT angiography on identifying vulnerable plaques compared to intravascular imaging | 1 day

SECONDARY OUTCOMES:
Overall coronary plaque detection rate using intravascular ultrasound as reference standard | 1 day
Total plaque volume | 1 day
minimum lumen area measurement compared to intravascular ultrasound | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Longjiang Zhang, MD, Study Chair — Jinling Hospital, Medical School of Nanjing University, Nanjing,China
Locations (1):
- Research Institute Of Medical Imaging Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Follmer B, Williams MC, Dey D, Arbab-Zadeh A, Maurovich-Horvat P, Volleberg RHJA, Rueckert D, Schnabel JA, Newby DE, Dweck MR, Guagliumi G, Falk V, Vazquez Mezquita AJ, Biavati F, Isgum I, Dewey M. Roadmap on the use of artificial intelligence for imaging of vulnerable atherosclerotic plaque in coronary arteries. Nat Rev Cardiol. 2024 Jan;21(1):51-64. doi: 10.1038/s41569-023-00900-3. Epub 2023 Jul 18. PMID 37464183
- [Background] Gaba P, Gersh BJ, Muller J, Narula J, Stone GW. Evolving concepts of the vulnerable atherosclerotic plaque and the vulnerable patient: implications for patient care and future research. Nat Rev Cardiol. 2023 Mar;20(3):181-196. doi: 10.1038/s41569-022-00769-8. Epub 2022 Sep 23. PMID 36151312
- [Result] Zhou F, Chen Q, Luo X, Cao W, Li Z, Zhang B, Schoepf UJ, Gill CE, Guo L, Gao H, Li Q, Shi Y, Tang T, Liu X, Wu H, Wang D, Xu F, Jin D, Huang S, Li H, Pan C, Gu H, Xie L, Wang X, Ye J, Jiang J, Zhao H, Fang X, Xu Y, Xing W, Li X, Yin X, Lu GM, Zhang LJ. Prognostic Value of Coronary CT Angiography-Derived Fractional Flow Reserve in Non-obstructive Coronary Artery Disease: A Prospective Multicenter Observational Study. Front Cardiovasc Med. 2022 Jan 31;8:778010. doi: 10.3389/fcvm.2021.778010. eCollection 2021. PMID 35174219